CLINICAL TRIAL: NCT06348316
Title: The Effect of Early Half Swaddling and Kangaroo Care Practices on Maternal Sleep Quality and Postpartum Depression in Term Babies: Randomized Controlled Study
Brief Title: Early Half Swaddling and Kangaroo Care Practices on Maternal Sleep Quality and Postpartum Depression in Term Babies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Burcu KUCUKKAYA, Principal Investigator, Trakya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TÜTF-GOBAEK 2023/45
Record Dates: First submitted 2024-03-30; First posted 2024-04-04 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Mothers; Postpartum Depression
Keywords: Term baby; Kangaroo care; Half swaddle; Sleep quality
MeSH Terms: conditions — Depression, Postpartum; Sleep Initiation and Maintenance Disorders | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention)
- Half swaddle (Experimental)
  Interventions: Other: Half swaddle
- Kangaroo care (Experimental)
  Interventions: Other: Kangaroo care
- Half swaddle+Kangaroo care (Experimental)
  Interventions: Other: Half swaddle; Other: Kangaroo care

INTERVENTIONS:
Other: Half swaddle — Half swaddle: HS applied to a newborn baby makes the baby feel completely safe, as if in the womb. After laying the soft fabric or baby blanket, it was placed in the supine position. Half swaddling was done so as not to restrict the baby's arm and leg movements. HS was performed 15 minutes before each sleep during the day until the 3rd month.
  Arms: Half swaddle; Half swaddle+Kangaroo care
Other: Kangaroo care — The application was applied twice a day and for 60 minutes every day for 6 months in a row. During KC, the mother placed her baby between two breasts, and the baby's breast was placed on the mother's breast in an upright position. During the application of KC, a quiet, calm, and the suitable environment was created so that comfort of the baby and mother would not be disturbed. The mother and baby are covered with a blanket. The ambient temperature was 26 centigrade degrees during the kangaroo care. In the continuation of the KB application, the mother was asked to breastfeed her baby. In order to prevent the risk of aspiration of the baby after breastfeeding, the baby was placed in the left lateral position so that the mother and the baby could lie down together. The researcher observed the application steps of the mother's KC, and the deficiencies, if any, were corrected by discussing with the mother during/after the application.
  Arms: Half swaddle+Kangaroo care; Kangaroo care

SUMMARY:
Aim: In this prospective, randomized controlled study, it was aimed to examine the effects of early half-swaddle and kangaroo care practices in term babies on maternal sleep quality and postpartum depression.

Design: The prospective, randomized controlled study

DETAILED DESCRIPTION:
The study will include n=136 mothers who gave birth at term at Trakya University Health Research and Application Center Birth Service. Between 10.09.2023 and 10.07.2024, n=136 (34=control, 34=semi-swaddled, 34=kangaroo care, 34=semi-swaddled and kangaroo care) women who volunteered to participate in the study will be conducted randomly in four groups: case and control.

Before starting the research, four groups will be randomly formed among the mothers. As a randomization method, mothers who meet the sampling inclusion criteria determined in the research will be identified and listed. Individuals to be taken into four groups will be determined by randomization method from the random numbers table. (http://www.stattrek.com/statistics/randomnumber-generator.aspx).

Research data: It was collected using the Survey Form, Edinburgh Postpartum Depression Scale (EPDS) and Pittsburgh Sleep Quality Index (PSQI).

Survey form; It which was prepared by the researchers by reviewing the literature consists of 5 main sections and a total of 82 questions, including the personal characteristics of the mother who gave birth preterm, the characteristics of the birth and the baby, the characteristics of sleep, the characteristics of the baby's sleep pattern, and the characteristics of the baby's growth and development.

Edinburgh Postnatal Depression Scale (EPDS): The scale was developed by Cox and Holden (1987). Adapted to Turkish by Engindeniz, Küey, and Kültür (1996). It is used to determine the risk for depression in the postnatal period and to measure the level and change of violence. It is a self-assessment scale. It is applied to postpartum women. It contains a total of 10 questions and measures depression. It provides a four-point Likert type measurement. The- Page 2 of 8 directive is at the beginning of the scale and subjects are asked to mark the substance most relevant to their situation when filling in the subjects. The total score of the scale is obtained by adding these item scores. As a result of the cut-off point scale study conducted in Turkey and it has ben calculated as 12/13.

Pittsburgh Sleep Quality Index (PSQI): PSQI is a self-reported screening and assessment questionnaire that details information on the type and severity of sleep quality and disorders within the last month. It was developed by Buysse et al., and its validity and reliability study in Turkish was performed by Agargün et al. PUKI evaluates sleep quality in the last month. 18 items and 7 components (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, daytime dysfunction) are included in the scoring. Each item is evaluated over 0-3 points and the sum of 7 component points gives the total PUKI score. The total score ranges from 0 to 21, with higher scores indicating worsening sleep quality. A total PUKI score of ≤5 is considered "good sleep", and >5 is considered "bad sleep".

The survey form and scales will be applied to all four groups at the first meeting. In the groups where half swaddle, kangaroo care and both half swaddle and kangaroo care are applied, necessary information about sleep, such as the mother's sleep duration, frequency of waking up, duration of wakefulness and reasons for waking up, will be recorded before the start of the study and for 24 hours. During the 6 months of the study period, mothers will be called every month by phone and their questions about the application methods and the application will be answered. All scales will be repeated at the beginning, 1st, 3rd and 6th months, and the mother's sleep monitoring for the last 24 hours will be requested again. Practical training on semi-swaddle and kangaroo care will be provided to mothers at the first meeting through prepared presentations.

Data collection The mean scores of PSQI and EPDS at the beginning,1st, 2nd, 3rd, and 6th months of the half swaddling and kangaroo care group Intervention.

Half swaddle: HS applied to a newborn baby makes the baby feel completely safe, as if in the womb. After laying the soft fabric or baby blanket, it was placed in the supine position. Half swaddling was done so as not to restrict the baby's arm and leg movements. HS was performed 15 minutes before each sleep during the day until the 3rd month.

Kangaroo care: The application was applied at twice a day and for 60 min, every day for 6 months in a row. While the mothers were taken to the NICU and practiced at home prior to kangaroo care, hand hygiene and breast care were provided within the scope of infection prevention rules. During KC, the mother placed her baby between two breasts, and the baby's breast was placed on the mother's breast in an upright position. During the application of KC, a quiet, calm and suitable environment was created so that comfort of the baby and mother would not be disturbed. The mother and baby are covered with a blanket. The ambient temperature was 26 centigrade degrees during the kangaroo care. In the continuation of the KB application, the mother was asked to breastfeed her baby. In order to prevent the risk of aspiration of the baby after breastfeeding, the baby was placed in the left lateral position so that the mother and the baby could lie down together. The application steps of the mother's KC were observed by the researcher and the deficiencies, if any, were corrected by discussing with the mother during / after the application.

Control group: The mothers in the control group were given routine care.

ELIGIBILITY:
Inclusion Criteria:

For mother;

* Over the age of 18-45,
* Term birth (single birth over 37 weeks),
* After an uncomplicated pregnancy, birth was completed by normal vaginal delivery or cesarean delivery method,
* Not using cigarettes, alcohol or stimulants,
* BMI<30,
* Not working night shifts,
* Having stable vital signs,
* Those who have not received infertility treatment,
* Does not have a chronic disease (such as hypertension, diabetes mellitus),
* Not experiencing serious depression, anxiety and stress,
* Does not have any organic or non-organic disease that may cause cognitive impairment (such as Delirium, Dementia, Mental Retardation, etc.),
* No serious maternal complications,
* Mothers who volunteer to participate in the research will be included in the study.

For baby;

* Having a birth weight above 2500 g,
* Having stable vital signs,
* Having an APGAR score above 7,
* No serious neonatal complications,
* Babies without congenital malformations will be included in the study.

Exclusion Criteria:

For mother;

* under 18 years old,
* Preterm birth (under 37 weeks and/or multiple birth),
* After a complicated pregnancy, birth has not been completed by normal vaginal delivery or cesarean delivery method,
* Those who use cigarettes, alcohol and stimulants,
* BMI>30,
* Working night shifts,
* Without stable vital signs,
* Those who have received infertility treatment,
* Having a chronic disease (such as hypertension, diabetes mellitus),
* Experiencing serious depression, anxiety and stress,
* Having any organic or non-organic disease that may cause cognitive impairment (such as Delirium, Dementia, Mental Retardation, etc.),
* Serious maternal complications,
* Mothers who do not volunteer to participate in the study will not be included in the study.

For baby;

* Birth weight of 2500 g or less,
* Without stable vital signs,
* Having an APGAR score below 7,
* Having serious neonatal complications,
* Babies with congenital malformations will not be included in the study.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2023-09-30 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Mother sleep quality evaluated using the Pittsburgh Sleep Quality Index (PSQI) | change from before implamentation patent and after 1st, 2nd, 3rd, and 6th months of practice.
  PSQI is a self-reported screening and assessment questionnaire that details information on the type and severity of sleep quality and disorders within the last month. It was developed by Buysse et al., and its validity and reliability study in Turkish was performed by Agargün et al. PUKI evaluates sleep quality in the last month. 18 items and 7 components (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, daytime dysfunction) are included in the scoring. Each item is evaluated over 0-3 points and the sum of 7 component points gives the total PUKI score. The total score ranges from 0 to 21, with higher scores indicating worsening sleep quality. A total PUKI score of ≤5 is considered "good sleep", and >5 is considered "bad sleep".
Postpartum depression evaluated using the Edinburgh Postnatal Depression Scale (EPDS) | change from before implamentation patent and after 1st, 2nd, 3rd, and 6th month of practice.
  The scale was developed by Cox and Holden (1987). Adapted to Turkish by Engindeniz, Küey, and Kültür (1996). It is used to determine the risk for depression in the postnatal period and to measure the level and change of violence. It is a self-assessment scale. It is applied to postpartum women. It contains a total of 10 questions and measures depression. It provides a four-point Likert type measurement. The directive is at the beginning of the scale and subjects are asked to mark the substance most relevant to their situation when filling in the subjects. The total score of the scale is obtained by adding these item scores. As a result of the cut-off point scale study conducted in Turkey and it has ben calculated as 12/13.

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Edirne, Turkey (Türkiye)

REFERENCES:
- [Derived] Kucukkaya B, Cihangir Ozturk T, Erginler G, Temiz M, Ercel O. The Effect of Early-Initiated Half-Swaddling and Kangaroo Care Practices on Maternal Sleep Quality and Postpartum Depression in Term Infants: A Randomized Controlled Trial. Nurs Health Sci. 2025 Mar;27(1):e70066. doi: 10.1111/nhs.70066. PMID 39988313